CLINICAL TRIAL: NCT06335758
Title: Non-randomized Observational Study to Collate Data Regarding the Safety, Efficacy and Satisfaction of ReX® in the Management of Solid Oral Medications.
Brief Title: Non-randomized Observational Study to Evaluate ReX® in the Management of Solid Oral Medication.
Acronym: RegStud
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dosentrx Ltd. (Industry)
Collaborators: US Oncology Research (Industry)
Responsible Party: Sponsor
Other Study IDs: EXC-039-2023-CLR
Record Dates: First submitted 2023-12-11; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-12

CONDITIONS: Any Solid Oral Medication
Keywords: Solid oral medication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving solid oral medication as a standard of care.: Solid oral medication administered via the ReX Remote Digital Nurse.
  Interventions: Device: Use of ReX to dispense and monitor solid oral medication therapy.

INTERVENTIONS:
Device: Use of ReX to dispense and monitor solid oral medication therapy. — ReX Remote Digital Nurse comprising hand-held dispenser, disposable drug cartridge and web application (ReX Treatment Manager).

SUMMARY:
The goal of this observational study is to evaluate the safety, efficacy and patient satisfaction with the ReX Remote Digital Nurse by patients receiving solid oral medication.

The study will evaluate and monitor use of ReX in respect of:

* treatment duration
* adverse events
* patient adherence and compliance
* engagement with ReX via patient-reported outcomes

Patients participating in the study will receive their normal medication as standard of care via ReX. Progress will be monitored via patients' responses to questions presented on the ReX touch screen.

DETAILED DESCRIPTION:
The ReX platform is a class 1 FDA device listed under product code NXB Dispenser Solid Medication. It comprises:

* Hand-held medication dispenser with touch screen (ReX Remote Digital Nurse).
* Disposable cartridge pre-loaded with pills or capsules. The cartridge includes an integral mouthpiece. Patients inhale at the mouthpiece causing pills to be dispensed into the mouth.
* Web application (ReX Treatment Manager) which collects data generated by the ReX hand-held dispenser.

ReX manages and monitors medication-based therapy by means of:

* Reminders to take pills. Reminders are sent to patients and caregivers by email, SMS or via the telephone support team.
* Electronic patient recorded outcomes (ePROs) presented to patients via the dispenser touch screen. ePROs include questions, tips and reminders.
* Notifications sent by email or SMS in the event of the patient exceeding a pre-defined threshold.

In this study, following training, patients will be offered their standard oral medication via the ReX Remote Digital Nurse. They will receive cartridges pre-loaded with medication by the pharmacy. Safety, efficacy and patient satisfaction with the device are monitored over a 24-week period by phone calls and periodic questionnaires.

Data collected by the ReX Remote Digital Nurse include:

* medication name
* prescribed dosage
* doses taken per day
* pills taken per dose
* ePRO responses
* missed pill intakes

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Care team recommends the use of ReX as a standard of care.
3. Patients have 5th grade reading level.
4. Patient was prescribed oral medication.
5. Patient takes medication at home.

Exclusion Criteria:

1. Patient has significant physical disability including poor fine motor skills, impaired visual or auditory faculties, mental disorders or other impairment affecting ability to provide Informed Consent or use the ReX dispensing unit effectively.
2. Patient failed to pass the learning module during ReX onboarding flow.
3. Patient is at end stage or terminal illness with anticipated life expectancy of 6 months or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive treatment with solid oral medication as a standard of care within ReX.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Treatment duration | 24 weeks
  At least 3 months while using ReX
Patient satisfaction | 24 weeks
  At least 3.5 on a scale up to 5
Adverse events | 24 weeks
  None related to use of ReX
Patient adherence | 24 weeks
  No. of pills taken by patient as a percentage of pills prescribed >80%
Patient compliance | 24 weeks
  No. of pills taken as percentage of pills to be taken in alloted time frame >70%
Patient engagement | 24 weeks
  No. of questions answered as a percentage of questions asked >70% of ePROs

CONTACTS AND LOCATIONS:
Overall Officials: David Waterhouse, MD, Principal Investigator — US Oncology
Locations (1):
- OHC, Cincinnati, Ohio, United States

REFERENCES:
- See also: Website of ReX Remote Digital Nurse — http://www.remotedigitalnurse.com